CLINICAL TRIAL: NCT05021458
Title: Comparison of Gong's Mobilization and Sustained Natural Apophyseal Glide on Pain and Range of Motion in Office Workers With Cervical Spine Overload
Brief Title: Gong's Mobilization and Sustained Natural Apophyseal Glide in Office Workers With Cervical Spine Overload
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/21/0113 Zaid
Record Dates: First submitted 2021-08-23; First posted 2021-08-25 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Cervical Spine Sprain
Keywords: mobilization,; cervical spine overload,; Gong's mobilization,; SNAGs

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Ten patients will be treated with Gong's mobilization.
  Interventions: Other: Gong's mobilization
- Group B (Active Comparator): Ten patients will be treated with SNAGs
  Interventions: Other: SNAG

INTERVENTIONS:
Other: Gong's mobilization — Ten patients will be treated with Gong's mobilization.
  Arms: Group A
Other: SNAG — : Ten patients will be treated with SNAGs
  Arms: Group B

SUMMARY:
Neck pain is a frequent and disabling complaint in the general population. One of the most common causes of neck pain is mechanical dysfunction of the cervical spine. Although diverse methods have been proposed for increasing cervical range of motion (ROM), joint mobilization has been confirmed as effective in several studies. Typically, joint mobilization methods for increasing cervical ROM include spinal manipulative therapy, the activator and diversified techniques. There are different mobilization techniques for neck pain, and mulligan's technique is one of them. It has two techniques Sustain Natural Apophyseal Glides (snags) and Natural Apophyseal Glides (nags). Gong's mobilization technique helps to heal physical pain as well as distract the mind from stress. In this study, the effectiveness of gong's mobilization and Sustained Natural Apophyseal Glides (snags) will be compared in office workers who have problems with cervical posture and range of motion (ROM) in order to examine the effects of gong's mobilization on cervical pain and cervical ROM. Twenty office workers with problems of cervical posture, pain and ROM is divided into a gong's mobilization group (n=10) and a Snags group (n=10). Gong's mobilization and nags will be administered three times a week for four weeks to each respective group and then changes in cervical posture, pain and cervical ROM will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* • Both Gender

  * Aged 25 to 45 years
  * Participants actively working in offices and who had been diagnosed with or self-reported chronic non-specific neck pain.
  * NPRS >4

Exclusion Criteria:

* • Surgical treatment of cervical spine (Cervical Diskectomy)

  * Tumor around the neck
  * Rheumatoid arthritis
  * Nervous system disorder(Vestibular disorder)
  * Whiplash Injury

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
universal Goniometer | 4 weeks
  range of joint
pain of patient | 4 weeks
  NPRS The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Function | 4 weeks
  Item scores range from 0 to 5, and the total score is a total of the item scores (possible range 0 (no pain) - 100 (maximal pain)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Salman Bashir, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gong W. The effects of cervical joint manipulation, based on passive motion analysis, on cervical lordosis, forward head posture, and cervical ROM in university students with abnormal posture of the cervical spine. J Phys Ther Sci. 2015 May;27(5):1609-11. doi: 10.1589/jpts.27.1609. Epub 2015 May 26. PMID 26157273
- [Background] Borghouts JAJ, Koes BW, Bouter LM. The clinical course and prognostic factors of non-specific neck pain: a systematic review. Pain. 1998 Jul;77(1):1-13. doi: 10.1016/S0304-3959(98)00058-X. PMID 9755013
- [Background] Jensen C. Development of neck and hand-wrist symptoms in relation to duration of computer use at work. Scand J Work Environ Health. 2003 Jun;29(3):197-205. doi: 10.5271/sjweh.722. PMID 12828389
- [Background] Cagnie B, Danneels L, Van Tiggelen D, De Loose V, Cambier D. Individual and work related risk factors for neck pain among office workers: a cross sectional study. Eur Spine J. 2007 May;16(5):679-86. doi: 10.1007/s00586-006-0269-7. Epub 2006 Dec 8. PMID 17160393